CLINICAL TRIAL: NCT00713232
Title: The Construction of a Chinese Picture Naming Test and Its Preliminary Normative Data
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Lu Lu, National Taiwan University Hospital
Other Study IDs: 200705052R
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2008-07-11 (Estimated); Status verified 2007-05

CONDITIONS: Normality
Keywords: naming test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- test construction: university student living in Taiwan for more than 5 years No known neurological, psychiatric or speech language disorders
- normative data: normal subjects 20-80 y/o Living in Taiwan for at least 5 years No know neurological, psychiatric and speech-language disorders

SUMMARY:
We will construct a Chinese Picture Naming test which include 60 items with various word frequency and familiarity and is arranged by their familiarity in daily life.

Then we will collect the normative data for this test using normal subjects of various age and educational level.

DETAILED DESCRIPTION:
In this study, we will first construct a Chinese Picture Naming Testing following the format of Boston Naming test. We will use the original 60 items from BNT and also choose another 100 items of objects with various frequency using the word frequency data from the Linguistic Corpus of the Academia Sinica. Colored pictures will be constructed accordingly. University students will be recruited to name the pictures and to judge the familiarity and image agreement for these pictures. Then, we will choose 60 pictures of according to the principles of 1. high image agreement 2. high naming agreement 3. including items of various familiarity and word frequency 4. double or triple phoneme words 5. including the original BNT items as possible. The 60 pictures will be arranged by their familiarity to construct the Chinese Picture Naming Test.

Then, we will recruit normal subjects of various age group and educational level to to the Naming test and to construct the preliminary norm.

ELIGIBILITY:
Inclusion Criteria:

* living in Taiwan for more than 5 years fluent in Chinese

Exclusion Criteria:

* previous neurological, psychiatric or speech language disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. university student
  2. normal subjects
Sampling Method: Non-Probability Sample
Enrollment: 522 (Actual)
Dates: Start 2007-05; Primary Completion 2007-06 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
naming accuracy | 10 minutes

SECONDARY OUTCOMES:
naming agreement | 10 min
image agreement | 10 min

CONTACTS AND LOCATIONS:
Overall Officials: Lu Lu, PhD, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan